CLINICAL TRIAL: NCT03487913
Title: A Phase 2, Open-Label, Multi-Center Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Lixivaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: The ELiSA Study - Evaluation of Lixivaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palladio Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-102
Record Dates: First submitted 2018-03-16; First posted 2018-04-04 (Actual); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — lixivaptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High dose lixivaptan / CKD1 or CKD2 (Experimental): Oral high dose lixivaptan in participants with CKD1 or CKD2
  Interventions: Drug: Lixivaptan
- Low dose lixivaptan / CKD1 or CKD2 (Experimental): Oral low dose lixivaptan in participants with CKD1 or CKD2
  Interventions: Drug: Lixivaptan
- High dose lixivaptan / CKD3 (Experimental): Oral high dose lixivaptan in participants with CKD3
  Interventions: Drug: Lixivaptan
- Low dose lixivaptan / CKD3 (Experimental): Oral low dose lixivaptan in participants with CKD3
  Interventions: Drug: Lixivaptan

INTERVENTIONS:
Drug: Lixivaptan — Oral vasopressin V2 receptor antagonist
  Other Names: VPA-985

SUMMARY:
This is a Phase 2, open-label, parallel-group, multiple dose study designed to evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of multiple doses of lixivaptan in Autosomal Dominant Polycystic Kidney Disease subjects with chronic kidney disease (CKD) in stages CKD1, CKD2 or CKD3.

DETAILED DESCRIPTION:
Therapeutic interventions aimed at counterbalancing the effect of vasopressin and/or normalizing intracellular levels of cAMP may be effective in delaying disease progression in autosomal dominant polycystic kidney disease (ADPKD).

The primary objectives of this study in subjects with ADPKD are:

* To characterize the safety and tolerability of lixivaptan following multiple doses in ADPKD subjects with relatively preserved kidney function (chronic kidney disease CKD1 and CKD2) and moderately impaired renal function (CKD3).

The secondary objectives of this study are:

* To characterize the PK profile of lixivaptan and its major metabolites following multiple doses of lixivaptan in ADPKD subjects with relatively preserved kidney function (CKD1 and CKD2) and moderately impaired renal function (CKD3).
* To characterize the pharmacodynamic effect of lixivaptan on urine output, urine osmolality, total kidney volume, serum vasopressin, and serum creatinine following multiple doses of lixivaptan in ADPKD subjects with relatively preserved kidney function (CKD1 and CKD2) and moderately impaired renal function (CKD3).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years of age at the time of screening
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 with eGFR calculated by the CKD EPI equation
* Diagnosed with ADPKD by modified Ravine criteria
* Considered by Investigator to be in good health relative to underlying CKD status and clinically stable with respect to underlying CKD

Exclusion Criteria:

* Known sensitivity or idiosyncratic reaction to lixivaptan, its related compounds such as benzazepines (e.g., tolvaptan, conivaptan, benazepril, fenoldopam, or mirtazapine), or any compound listed as being present in the study formulation
* Women who are pregnant or breast feeding
* Subjects have taken tolvaptan, oral or intravenous antibiotics, or any investigational drug or used an investigational device within 30 days or 5 half-lives, whichever is longer, prior to first study dose
* Subject has a transplanted kidney, or absence of a kidney
* Subjects with clinically significant incontinence, overactive bladder, or urinary retention (e.g., benign prostatic hyperplasia)
* Subjects with clinically significant liver disease, or clinically significant liver function abnormalities or serology other than that expected for ADPKD with cystic liver disease at baseline
* Subjects with any clinically significant concomitant disease or condition other than ADPKD (including treatment for such conditions) that, in the opinion of the Investigator, could either interfere with the study drug or pose an unacceptable risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente E Torres, MD, PhD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (12):
  - Palladio Biosciences Clinical Site, Los Angeles, California
  - Palladio Biosciences Clinical Site, Jacksonville, Florida
  - Palladio Biosciences Clinical Site, Miami, Florida
  - Palladio Biosciences Clinical Site, Palmetto Bay, Florida
  - Palladio Biosciences Clinical Site, Tampa, Florida
  - Palladio Biosciences Clinical Site, Baltimore, Maryland
  - Palladio Biosciences Clinical Site, Rochester, Minnesota
  - Palladio Biosciences Clinical Site, Kansas City, Missouri
  - Palladio Biosciences Clinical Site, Laurelton, New York
  - Palladio Biosciences Clinical Site, Indiana, Pennsylvania
  - Palladio Biosciences Clinical Site, Nashville, Tennessee
  - Palladio Biosciences Clinical Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shusterman NH, Hogan LC, Pellegrini L: Effect of lixivaptan on pharmacokinetic (PK) and pharmacodynamic (PD) end points in patients with autosomal dominant polycystic kidney disease (ADPKD) in the ELiSA Study (PA-102) [Abstract]. J Am Soc Nephrol 30, 2019 (abstract supplement issue): page 339.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Started | 9 | 7 | 8 | 7
Completed | 9 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3 | Total
Number analyzed (Participants) | 9 | 7 | 8 | 7 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 8 | 7 | 31
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (16.99) | 34.9 (10.85) | 54.0 (9.07) | 51.6 (10.54) | 45.1 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 4 | 18
  Male | 4 | 2 | 4 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 2 | 8
  Not Hispanic or Latino | 9 | 5 | 4 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 7 | 8 | 7 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter Cmax, the highest concentration of lixivaptan measured in plasma after multiple doses of drug, will be calculated from the observed concentration of lixivaptan and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Of these, all 31 subjects contributed to the PK data on Day 1 (am); 30 contributed data to Day 1 (pm); and 29 contributed data to Day 7 (am) and (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng/mL
  Day 1 (am) | 656.8 (28.1) | 190.9 (52.0) | 681.3 (45.9) | 156.9 (66.9)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 1007 (36.6) | 211.5 (33.5) | 930.2 (44.5) | 159.5 (51.9)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 1442 (34.3) | 339.5 (19.5) | 1422 (48.3) | 276.9 (33.7)
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 1582 (45.8) | 301.0 (13.7) | 1211 (90.5) | 258.8 (38.4)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter Cmax, the highest concentration of WAY-141624 measured in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-141624 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Missing values and substantial deviations from planned dosing interval durations meant results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng/mL
  Day 1 (am): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (am) | 455.3 (33.3) | 123.7 (69.7) | 381.7 (46.6) | 135.3 (55.5)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 561.7 (35.4) | 160.8 (56.0) | 417.8 (41.4) | 142.3 (28.7)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 535.8 (34.4) | 213.8 (75.4) | 652.1 (49.0) | 233.7 (50.8)
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 612.6 (42.3) | 200.1 (63.0) | 588.5 (69.2) | 224.8 (44.7)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter Cmax, the highest concentration of WAY-138451 measured in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-138451 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Missing values, substantial deviations, and <3 quantifiable postdose WAY-138451 concentrations meant results were excluded from subjects at various time points.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng/mL
  Day 1 (am): number analyzed (Participants) | 9 | 4 | 8 | 5
  Day 1 (am) | 84.33 (28.3) | 28.83 (21.4) | 82.23 (56.3) | 24.74 (38.6)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 6
  Day 1 (pm) | 117.1 (38.1) | 25.93 (25.4) | 103.3 (38.3) | 20.95 (35.4)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 177.4 (22.8) | 40.79 (27.6) | 165.4 (43.1) | 33.61 (36.2)
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 189.1 (35.2) | 35.36 (10.4) | 155.2 (74.0) | 31.64 (20.2)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter Cmax, the highest concentration of WAY-138758 measured in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-138758 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Of these, all 31 subjects contributed to the PK data on Day 1 (am); 30 contributed data to Day 1 (pm); and 29 contributed data to Day 7 (am) and (pm). Substantial deviations from planned dosing interval durations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng/mL
  Day 1 (am) | 239.3 (40.3) | 85.11 (36.5) | 185.2 (49.7) | 64.26 (53.9)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 354.6 (32.8) | 125.5 (53.8) | 275.0 (26.5) | 107.1 (43.5)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 822.3 (54.4) | 320.4 (60.4) | 833.6 (25.0) | 343.9 (35.8)
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 861.4 (56.0) | 326.8 (56.7) | 825.2 (24.0) | 342.2 (36.0)

5. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter tmax, the time taken to reach the highest concentration of lixivaptan in plasma after multiple doses of drug, will be calculated from the observed concentration of lixivaptan and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Of these, all 31 subjects contributed to the PK data on Day 1 (am); 30 contributed data to Day 1 (pm); and 29 contributed data to Day 7 (am) and (pm). Substantial deviations from planned dosing interval durations meant results were excluded from subjects at various time points.
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am) | 1.000 [1.00 to 1.00] | 1.000 [1.00 to 1.05] | 1.000 [1.00 to 2.00] | 1.020 [0.67 to 2.00]
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 1.000 [0.97 to 2.00] | 1.000 [1.00 to 1.93] | 1.000 [1.00 to 5.97] | 0.980 [0.95 to 5.62]
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 1.000 [1.00 to 1.00] | 1.000 [1.00 to 1.02] | 1.000 [1.00 to 2.00] | 1.000 [0.78 to 1.05]
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 1.000 [1.00 to 2.00] | 1.000 [0.95 to 1.03] | 1.000 [0.97 to 13.95] | 0.920 [0.83 to 1.67]

6. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter tmax, the time taken to reach the highest concentration of WAY-141624 in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-141624 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (am) | 2.000 [1.00 to 4.00] | 2.000 [1.05 to 2.00] | 2.000 [1.00 to 4.00] | 2.000 [1.67 to 4.00]
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 2.000 [2.00 to 4.00] | 2.000 [1.93 to 4.03] | 2.000 [0.00 to 4.00] | 1.950 [1.92 to 13.58]
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 2.000 [1.00 to 2.00] | 2.000 [2.00 to 2.03] | 2.000 [1.00 to 4.08] | 2.000 [1.83 to 2.00]
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 2.000 [2.00 to 4.00] | 2.010 [1.93 to 5.95] | 2.025 [0.00 to 13.95] | 1.920 [1.67 to 2.00]

7. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter tmax, the time taken to reach the highest concentration of WAY-138451 in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-138451 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. Missing values, substantial deviations from planned dosing interval durations, and <3 quantifiable postdose WAY-138451 concentrations meant results were excluded from subjects at various time points.
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 9 | 4 | 8 | 5
  Day 1 (am) | 1.000 [1.00 to 2.00] | 1.010 [1.00 to 1.05] | 1.000 [1.00 to 2.00] | 1.020 [0.67 to 2.00]
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 6
  Day 1 (pm) | 1.000 [0.97 to 2.00] | 1.475 [1.00 to 2.00] | 2.000 [0.92 to 5.97] | 0.975 [0.95 to 1.93]
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 1.000 [1.00 to 1.00] | 1.000 [1.00 to 2.00] | 2.000 [1.00 to 2.08] | 1.050 [0.95 to 2.00]
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 1.000 [1.00 to 2.00] | 1.015 [1.00 to 1.95] | 3.000 [1.00 to 13.95] | 1.000 [0.83 to 2.00]

8. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter tmax, the time taken to reach the highest concentration of WAY-138758 in plasma after multiple doses of drug, will be calculated from the observed concentration of WAY-138758 and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. All 31 subjects in the PKAS contributed to the PK data on Day 1 (am); 30 contributed data to Day 1 (pm); and 29 contributed data to Day 7 (am) and (pm). Substantial deviations from planned dosing interval durations and missing values meant results were excluded from subjects at various time points.
Measure: Median (Full Range); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am) | 4.000 [2.00 to 6.00] | 4.030 [4.00 to 6.00] | 9.460 [6.00 to 10.00] | 4.020 [3.68 to 9.93]
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 4.000 [2.00 to 13.87] | 4.000 [2.00 to 13.83] | 4.000 [4.00 to 13.95] | 13.400 [3.98 to 13.87]
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 4.000 [0.00 to 6.00] | 2.030 [2.00 to 4.00] | 3.000 [0.00 to 9.92] | 5.980 [0.00 to 9.75]
  Day 7 (pm): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (pm) | 2.000 [1.00 to 13.98] | 3.010 [2.00 to 6.10] | 4.000 [0.00 to 13.95] | 3.900 [0.00 to 5.97]

9. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until the Last Quantifiable Concentration (AUC[0-last]) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-last) for lixivaptan will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values, summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: The PKAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan, underwent plasma PK sampling, and were evaluable for this PK outcome. All 31 subjects in the PKAS contributed to the PK data on Day 1 (am); 30 contributed data to Day 1 (pm); 29 contributed data to Day 7 (am), and 27 contributed data to Day 7 (pm). Substantial deviations from planned dosing interval durations and missing values meant results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng*hour/mL
  Day 1 (am) | 1688 (43.5) | 506.7 (45.0) | 2281 (37.9) | 428.8 (46.6)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 3619 (48.5) | 782.1 (15.7) | 5208 (46.3) | 782.8 (24.7)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 4237 (36.8) | 1007 (27.7) | 5395 (35.3) | 889.4 (29.7)
  Day 7 (pm): number analyzed (Participants) | 7 | 5 | 8 | 7
  Day 7 (pm) | 8467 (47.2) | 1958 (80.2) | 12870 (56.2) | 1666 (56.0)

10. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until the Last Quantifiable Concentration (AUC[0-last]) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-last) for WAY-141624 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng*hour/mL
  Day 1 (am): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (am) | 2339 (44.1) | 669.1 (48.8) | 2300 (43.1) | 716.5 (54.2)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 3963 (48.7) | 1214 (49.3) | 3894 (29.0) | 1266 (45.7)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 3440 (40.4) | 1349 (58.1) | 4196 (37.7) | 1560 (56.9)
  Day 7 (pm): number analyzed (Participants) | 7 | 6 | 8 | 7
  Day 7 (pm) | 11330 (56.4) | 4174 (56.3) | 15160 (54.8) | 4731 (81.2)

11. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until the Last Quantifiable Concentration (AUC[0-last]) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-last) for WAY-138451 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng*hour/mL
  Day 1 (am): number analyzed (Participants) | 9 | 4 | 8 | 5
  Day 1 (am) | 284.7 (50.3) | 77.23 (24.8) | 373.6 (44.9) | 70.01 (21.6)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 6
  Day 1 (pm) | 532.8 (65.5) | 80.14 (36.1) | 764.5 (40.1) | 74.00 (26.9)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 736.8 (31.2) | 139.7 (45.1) | 919.2 (39.8) | 132.9 (42.4)
  Day 7 (pm): number analyzed (Participants) | 6 | 5 | 8 | 7
  Day 7 (pm) | 1444 (52.6) | 194.6 (138.3) | 1867 (58.8) | 137.3 (46.5)

12. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until the Last Quantifiable Concentration (AUC[0-last]) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-last) for WAY-138758 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values and summarized by cohort.
Time Frame: Day 1 (am and pm) and Day 7 (am and pm)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
ng*hour/mL
  Day 1 (am) | 1792 (36.9) | 669.7 (37.1) | 1412 (51.3) | 485.1 (65.0)
  Day 1 (pm): number analyzed (Participants) | 9 | 6 | 8 | 7
  Day 1 (pm) | 4281 (35.3) | 1449 (50.7) | 3418 (24.5) | 1212 (49.2)
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 7471 (54.5) | 2919 (59.2) | 7660 (24.6) | 3162 (36.3)
  Day 7 (pm): number analyzed (Participants) | 7 | 6 | 8 | 7
  Day 7 (pm) | 46910 (62.8) | 18940 (51.9) | 52560 (28.0) | 23890 (38.1)

13. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf]) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-inf) for lixivaptan will be calculated using the linear trapezoidal rule for increasing values, the log trapezoidal rule for decreasing values, and extrapolated to infinity by addition of the last quantifiable observed concentration divided by the elimination rate constant and summarized by cohort.
Time Frame: Day 1 (am)
Population: Upon final PK data analysis, it was evident based upon Day 7 PM profiles (sampled out to 96 hours) that lixivaptan did not appear to have concentration-time data in the terminal phase for Day 1 (AM) or Day 7 AM due to the limited time frame of the dosing intervals of 10 hours. Therefore, the terminal slope-related PK parameter of AUC(0-inf), planned in the protocol/SAP for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose.
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf]) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-inf) for WAY-141624 will be calculated using the linear trapezoidal rule for increasing values, the log trapezoidal rule for decreasing values, and extrapolated to infinity by addition of the last quantifiable observed concentration divided by the elimination rate constant and summarized by cohort.
Time Frame: Day 1 (am)
Population: Upon final PK data analysis, it was evident based upon Day 7 PM profiles (sampled out to 96 hours) that WAY-141624 did not appear to have concentration-time data in the terminal phase for Day 1 (AM) or Day 7 AM due to the limited time frame of the dosing intervals of 10 hours. Therefore, the terminal slope-related PK parameter of AUC(0-inf), planned in the protocol/SAP for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose.
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf]) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-inf) for WAY-138451 will be calculated using the linear trapezoidal rule for increasing values, the log trapezoidal rule for decreasing values, and extrapolated to infinity by addition of the last quantifiable observed concentration divided by the elimination rate constant and summarized by cohort.
Time Frame: Day 1 (am)
Population: Upon final PK data analysis, it was evident based upon Day 7 PM profiles (sampled out to 96 hours) that WAY-138451 did not appear to have concentration-time data in the terminal phase for Day 1 (AM) or Day 7 AM due to the limited time frame of the dosing intervals of 10 hours. Therefore, the terminal slope-related PK parameter of AUC(0-inf), planned in the protocol/SAP for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose.
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf]) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-inf) for WAY-138758 will be calculated using the linear trapezoidal rule for increasing values, the log trapezoidal rule for decreasing values, and extrapolated to infinity by addition of the last quantifiable observed concentration divided by the elimination rate constant and summarized by cohort.
Time Frame: Day 1 (am)
Population: Upon final PK data analysis, it was evident based upon Day 7 PM profiles (sampled out to 96 hours) that WAY-138758 did not appear to have concentration-time data in the terminal phase for Day 1 (AM) or Day 7 AM due to the limited time frame of the dosing intervals of 10 hours. Therefore, the terminal slope-related PK parameter of AUC(0-inf), planned in the protocol/SAP for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose.
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Primary Outcome: Terminal Elimination Phase Half-life (t1/2) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter t1/2 for lixivaptan, determined as ln2/apparent terminal elimination rate constant, will be calculated and summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that lixivaptan did not have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, t1/2, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values and substantial deviations meant results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 6 | 4 | 7 | 6
  Day 7 (pm) | 9.696 (24.2) | 7.688 (51.6) | 11.39 (28.9) | 10.25 (27.4)

18. Primary Outcome: Terminal Elimination Phase Half-life (t1/2) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter t1/2 for WAY-141624, determined as ln2/apparent terminal elimination rate constant, will be calculated and summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that WAY-141624 did not have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, t1/2, planned for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values and substantial deviations meant results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 7 | 4 | 8 | 5
  Day 7 (pm) | 20.48 (33.3) | 22.41 (56.1) | 20.81 (30.4) | 18.79 (22.2)

19. Primary Outcome: Terminal Elimination Phase Half-life (t1/2) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter t1/2 for WAY-138451, determined as ln2/apparent terminal elimination rate constant, will be calculated and summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: It was evident WAY-138451 did not have concentration-time data in the terminal phase for D1(am) due to the limited time frame of the 10-hour dosing intervals. t1/2, planned for Day 1 AM, was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values, substantial deviations and <3 quantifiable postdose WAY-138451 concentrations meant some results were excluded; also, t1/2 could not be calculated for the 2 participants in the low dose lixivaptan/CKD3 cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 7 | 0 | 6 | 2
  Day 7 (pm) | 6.439 (36.7) |  | 9.426 (22.6) | NA (NA) — Insufficient number of subjects with data to calculate the geometric mean

20. Primary Outcome: Terminal Elimination Phase Half-life (t1/2) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter t1/2 for WAY-138758, determined as ln2/apparent terminal elimination rate constant, will be calculated and summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that WAY-138758 did not appear to have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, t1/2, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
hours
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 8 | 5 | 8 | 6
  Day 7 (pm) | 48.80 (25.8) | 50.70 (8.6) | 59.93 (32.8) | 65.11 (30.2)

21. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter λZ for lixivaptan will be determined by linear regression of the terminal points of the log-linear concentration-time curve. The Best Fit method utilized by WinNonlin will be used to identify the terminal linear phase of the concentration-time profile, with visual assessment and adjustment of the selected data points by the PK scientist if warranted. A minimum of 3 data points will be used for determination. Results will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that lixivaptan did not appear to have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, λZ, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
1/hour
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 6 | 4 | 7 | 6
  Day 7 (pm) | 0.07149 (24.2) | 0.09016 (51.6) | 0.06085 (28.9) | 0.06762 (27.4)

22. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter λZ for WAY-141624 will be determined by linear regression of the terminal points of the log-linear concentration-time curve. The Best Fit method utilized by WinNonlin will be used to identify the terminal linear phase of the concentration-time profile, with visual assessment and adjustment of the selected data points by the PK scientist if warranted. A minimum of 3 data points will be used for determination. Results will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that WAY-141624 did not appear to have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, λZ, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the PM dose. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
1/hour
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 7 | 4 | 8 | 5
  Day 7 (pm) | 0.03384 (33.3) | 0.03093 (56.1) | 0.03330 (30.4) | 0.03690 (22.2)

23. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter λZ for WAY-138451 will be determined by linear regression of the terminal points of the log-linear concentration-time curve. The Best Fit method utilized by WinNonlin will be used to identify the terminal linear phase of the concentration-time profile, with visual assessment and adjustment of the selected data points by the PK scientist if warranted. A minimum of 3 data points will be used for determination. Results will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: It was evident WAY-138451 did not appear to have concentration-time data in the terminal phase for D1(am) due to the limited time frame of the dosing intervals of 10 hours. λZ, planned for D1(am), was unable to be calculated due to insufficient sampling duration prior to the pm dose. Missing values, deviations, and <3 quantifiable postdose WAY-138451 concentrations meant results were excluded; also, λZ could not be calculated for the 2 participants in the low dose lixivaptan/CKD3 cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
1/hour
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 7 | 0 | 6 | 2
  Day 7 (pm) | 0.1077 (36.7) |  | 0.07353 (22.6) | NA (NA) — Insufficient number of subjects with data to calculate the geometric mean

24. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter λZ for WAY-138758 will be determined by linear regression of the terminal points of the log-linear concentration-time curve. The Best Fit method utilized by WinNonlin will be used to identify the terminal linear phase of the concentration-time profile, with visual assessment and adjustment of the selected data points by the PK scientist if warranted. A minimum of 3 data points will be used for determination. Results will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (pm)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that WAY-138758 did not appear to have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, λZ, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the pm dose. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
1/hour
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (pm): number analyzed (Participants) | 8 | 5 | 8 | 6
  Day 7 (pm) | 0.01421 (25.8) | 0.01367 (8.6) | 0.01157 (32.8) | 0.01065 (30.2)

25. Primary Outcome: Apparent Systemic Clearance After Extravascular Dosing (CL/F) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter CL/F for lixivaptan, calculated as: Day 1 AM: dose divided by AUC(0-inf), or Day 7 AM: dose divided by AUC(0-last), will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (am)
Population: Upon final PK data analysis, it was evident based upon Day 7 (pm) profiles that lixivaptan did not appear to have concentration-time data in the terminal phase for Day 1 (am) due to the limited time frame of the dosing intervals of 10 hours. Therefore, CL/F, planned for Day 1 (am), was unable to be calculated due to insufficient sampling duration prior to the pm dose. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
L/hour
  Day 1 (am): number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 7 (am): number analyzed (Participants) | 8 | 6 | 8 | 7
  Day 7 (am) | 47.20 (36.8) | 49.65 (27.7) | 37.07 (35.3) | 56.22 (29.7)

26. Primary Outcome: Volume of Distribution After Extravascular Dosing (VZ/F) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter VZ/F for lixivaptan, calculated as CL/F divided by λZ, will be summarized by cohort.
Time Frame: Day 1 (am) and Day 7 (am)
Population: Upon final data analysis, it was evident based upon Day (D) 7(pm) profiles that lixivaptan did not have concentration-time data in the terminal phase for D1(am) due to the limited time frame of the 10-hour dosing intervals. Therefore, VZ/F, planned for D1(am), was unable to be calculated due to insufficient sampling duration prior to the pm dose, and values for the D7(am) time point were not presented. Instead, VZ/F24H was determined and presented as an Other Pre-specified Outcome Measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7

27. Primary Outcome: Accumulation Ratio for Cmax (RCmax) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter RCmax for lixivaptan, calculated as [Cmax on Day 7]/[Cmax on Day 1], will be summarized by cohort.
Time Frame: Day 7 (am)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (am).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 2.287 (24.1) | 1.687 (68.4) | 2.087 (36.2) | 1.765 (50.1)

28. Primary Outcome: Accumulation Ratio for AUC(0-last) (RAUC[0-last]) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter RAUC(0-last) for lixivaptan, calculated as [AUC(0-last) on Day 7]/[AUC(0-last) on Day 1], will be summarized by cohort.
Time Frame: Day 7 (am)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (am).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 2.643 (28.6) | 1.795 (25.6) | 2.365 (28.9) | 2.074 (31.5)

29. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until 14 Hours Postdose (AUC[0-14]) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-14) for lixivaptan will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values. The actual elapsed time for the nominal 14-hour sample will be used for the calculation. Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
ng*h/mL | 6530 (44.3) | 1280 (26.9) | 7800 (55.2) | 1069 (29.0)

30. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until 14 Hours Postdose (AUC[0-14]) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-14) for WAY-141624 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values. The actual elapsed time for the nominal 14-hour sample will be used for the calculation. Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
ng*h/mL | 5227 (46.6) | 1717 (46.6) | 5871 (50.7) | 1959 (54.0)

31. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until 14 Hours Postdose (AUC[0-14]) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-14) for WAY-138451 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values. The actual elapsed time for the nominal 14-hour sample will be used for the calculation. Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
ng*h/mL | 1107 (39.2) | 182.8 (33.4) | 1270 (50.8) | 154.4 (37.7)

32. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Until 14 Hours Postdose (AUC[0-14]) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter AUC(0-14) for WAY-138758 will be calculated using the linear trapezoidal rule for increasing values and the log trapezoidal rule for decreasing values. The actual elapsed time for the nominal 14-hour sample will be used for the calculation. Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
ng*h/mL | 10900 (55.6) | 4121 (56.9) | 10730 (25.3) | 4509 (36.2)

33. Primary Outcome: Ratio of WAY-141624 Cmax to Parent Lixivaptan Cmax (MRCmax) in ADPKD Patients
Description: The pharmacokinetic parameter MRCmax for WAY-141624 will be calculated and corrected for molecular weight of WAY-141624 and parent lixivaptan as: (Cmax,m/Cmax,p)(MWp/MWm), where Cmax,m and MWm are Cmax and molecular weight of WAY-141624, respectively, and Cmax,p and MWp are Cmax and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRCmax calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-141624: 505.95 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 0.3627 (40.0) | 0.6225 (57.5) | 0.4554 (31.0) | 0.8137 (41.5)

34. Primary Outcome: Ratio of WAY-138451 Cmax to Parent Lixivaptan Cmax (MRCmax) in ADPKD Patients
Description: The pharmacokinetic parameter MRCmax for WAY-138451 will be calculated and corrected for molecular weight of WAY-138451 and parent lixivaptan as: (Cmax,m/Cmax,p)(MWp/MWm), where Cmax,m and MWm are Cmax and molecular weight of WAY-138451, respectively, and Cmax,p and MWp are Cmax and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRCmax calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-138451: 488.92 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 0.1159 (17.7) | 0.1139 (14.9) | 0.1243 (27.5) | 0.1185 (29.3)

35. Primary Outcome: Ratio of WAY-138758 Cmax to Parent Lixivaptan Cmax (MRCmax) in ADPKD Patients
Description: The pharmacokinetic parameter MRCmax for WAY-138758 will be calculated and corrected for molecular weight of WAY-138758 and parent lixivaptan as: (Cmax,m/Cmax,p)(MWp/MWm), where Cmax,m and MWm are Cmax and molecular weight of WAY-138758, respectively, and Cmax,p and MWp are Cmax and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRCmax calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-138758: 426.82 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 0.6045 (61.7) | 1.205 (56.9) | 0.7569 (86.0) | 1.468 (51.2)

36. Primary Outcome: Ratio of Metabolite AUC(0-14) to Parent Lixivaptan AUC(0-14) (MRAUC[0-14]) of WAY-141624 in ADPKD Patients
Description: The pharmacokinetic parameter MRAUC(0-14) for WAY-141624 will be calculated and corrected for molecular weight of WAY-141624 and parent lixivaptan as: (AUC(0-14),m/AUC(0-14),p)(MWp/MWm), where AUC(0-14),m and MWm are AUC(0-14) and molecular weight of WAY-141624, respectively, and AUC(0-14),p and MWp are AUC(0-14) and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRAUC(0-14) calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-141624: 505.95 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 0.7498 (41.0) | 1.256 (69.7) | 0.7050 (24.1) | 1.717 (42.7)

37. Primary Outcome: Ratio of Metabolite AUC(0-14) to Parent Lixivaptan AUC(0-14) (MRAUC[0-14]) of WAY-138451 in ADPKD Patients
Description: The pharmacokinetic parameter MRAUC(0-14) for WAY-138451 will be calculated and corrected for molecular weight of WAY-138451 and parent lixivaptan as: (AUC(0-14),m/AUC(0-14),p)(MWp/MWm), where AUC(0-14),m and MWm are AUC(0-14) and molecular weight of WAY-138451, respectively, and AUC(0-14),p and MWp are AUC(0-14) and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRAUC(0-14) calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-138451: 488.92 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 0.1643 (10.9) | 0.1384 (11.3) | 0.1579 (17.5) | 0.1401 (23.9)

38. Primary Outcome: Ratio of Metabolite AUC(0-14) to Parent Lixivaptan AUC(0-14) (MRAUC[0-14]) of WAY-138758 in ADPKD Patients
Description: The pharmacokinetic parameter MRAUC(0-14) for WAY-138758 will be calculated and corrected for molecular weight of WAY-138758 and parent lixivaptan as: (AUC(0-14),m/AUC(0-14),p)(MWp/MWm), where AUC(0-14),m and MWm are AUC(0-14) and molecular weight of WAY-138758, respectively, and AUC(0-14),p and MWp are AUC(0-14) and molecular weight of parent lixivaptan, respectively. The following molecular weights are to be used in all MRAUC(0-14) calculations:
  * lixivaptan: 473.93 g/mol
  * WAY-138758: 426.82 g/mol
  Results will be summarized by cohort.
Time Frame: Day 7 (pm)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (pm).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 8 | 6 | 8 | 7
Ratio | 1.854 (64.2) | 3.573 (83.1) | 1.528 (53.7) | 4.685 (39.7)

39. Primary Outcome: Number of Study Participants With Treatment-emergent Adverse Events
Description: The number of study participants who experience treatment-emergent adverse events during the study will be counted and summarized by dose level.
Time Frame: 35 days
Population: Results are presented based on the Safety Analysis Set, which included all subjects who received at least 1 dose of study medication, and were analyzed according to treatment received. The Safety Analysis Set included all 31 subjects who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants | 2 | 4 | 4 | 4

40. Primary Outcome: Number of Study Participants With Clinically Significant Physical Examination Findings
Description: The number of study participants who experience clinically significant physical examination findings during the study will be counted and summarized by cohort.
Time Frame: 35 days
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants | 0 | 0 | 0 | 1

41. Primary Outcome: Number of Study Participants With Clinically Significant Vital Signs
Description: The number of study participants who experience vital signs (systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, and body temperature) meeting the predefined markedly abnormal criteria during the study will be counted and summarized by cohort.
Time Frame: 35 days
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants | 0 | 0 | 0 | 0

42. Primary Outcome: Number of Study Participants With Clinically Significant Changes in 12-lead Electrocardiograms
Description: The number of study participants who experience 12-lead electrocardiograms meeting the predefined markedly abnormal criteria during the study will be counted and summarized by cohort.
Time Frame: Baseline (Day 1) to Day 8 (8 days)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants | 0 | 0 | 0 | 0

43. Primary Outcome: Number of Study Participants With Abnormal Clinical Laboratory Findings (Including Clinical Chemistry, Hematology, and Urinalysis)
Description: The number of study participants who experience clinically meaningful laboratory findings, relating to clinical chemistry, hematology, and urinalysis, during the study will be counted and summarized by cohort.
Time Frame: 35 days
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants
  Clinical chemistry | 0 | 0 | 0 | 0
  Hematology | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0

44. Primary Outcome: Aquaretic Tolerability of Lixivaptan Measured by a Tolerability Questionnaire Relating to the Symptom Burden of Nocturia, Urgency, and Frequency at Day 7: Questions 1, 2, 6, and 10
Description: The number of study participants who answered "yes" to the following questions at Day 7 will be counted and summarized by dose level:
  * Could you tolerate taking this dose of study drug for the next 12 months?
  * Did the study drug make you feel thirsty more often than usual?
  * Did the study drug make you go to the bathroom (urinate) more often than usual during the night?
  * Would you be comfortable recommending the study drug to another patient with your kidney condition?
Time Frame: Day 7
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
Participants
  Could you tolerate taking this dose of study drug for the next 12 months? | 7 | 6 | 7 | 7
  Did the study drug make you feel thirsty more often than usual? | 7 | 6 | 8 | 4
  Did the study drug make you go to the bathroom (urinate) more often than usual during the night? | 6 | 3 | 6 | 4
  Would you be comfortable recommending the study drug to another patient with your kidney condition? | 9 | 7 | 8 | 7

45. Primary Outcome: Aquaretic Tolerability of Lixivaptan Measured by a Tolerability Questionnaire Relating to the Symptom Burden of Nocturia, Urgency, and Frequency at Day 7: Question 3
Description: The number of study participants who answered "not at all" and "slightly" to the following question at Day 7 will be measured:
  • If the study drug made you feel thirsty more often than usual, were you bothered by it?
Time Frame: Day 7
Population: Results are presented based on the Safety Analysis Set, which included all subjects who received at least 1 dose of study medication, and were analyzed according to treatment received. The Safety Analysis Set included all 31 subjects who were enrolled in the study. Answers were not received from all participants.
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose Lixivaptan / CKD1 or CKD2; High Dose Lixivaptan / CKD3; Low Dose Lixivaptan / CKD3: Oral high dose lixivaptan in participants with CKD1 or CKD2
  Lixivaptan: Oral vasopressin V2 receptor antagonist
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 7 | 6 | 8 | 4
Participants
  Answered "not at all" | 2 | 2 | 4 | 2
  Answered "slightly" | 4 | 2 | 3 | 0

46. Secondary Outcome: Change From Baseline in Spot Urine Osmolality
Description: Changes from baseline in spot urine measurements for samples taken at 0, 1, 2, 4, 6, 9, 10, 11, 12, 14, and 24 hours after the Day 1 and Day 7 doses will be summarized by cohort. The baseline value for each time point after first administration of study drug is the value observed at the corresponding time point on Day -1 (or Day 1 for the AM predose assessment only).
Time Frame: At time of dose, and at 1, 2, 4, 6, 9, 10, 11, 12, 14, and 24 hours after the Day 1 and Day 7 doses
Population: The Pharmacodynamic Analysis Set (PDAS) consisted of all 31 subjects in the Safety analysis set who received lixivaptan. Overall, all 31 subjects contributed PD endpoints to the Day 1/2 assessment; 30 subjects contributed data to the Day 7/8 PD endpoints and scheduled EOS assessments; however, values were not available for all participants at each time point.
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mOsm/kg
  Time of Day 1 dose: number analyzed (Participants) | 9 | 7 | 6 | 7
  Time of Day 1 dose | -27.7 (253.8) | -28.4 (183.5) | -52.3 (56.1) | -167.3 (63.4)
  1 hour post Day 1 dose: number analyzed (Participants) | 9 | 7 | 6 | 7
  1 hour post Day 1 dose | -101.9 (150.2) | 6.1 (60.1) | -44.2 (68.7) | -114.7 (95.0)
  2 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  2 hours post Day 1 dose | -10.1 (25.1) | -41.6 (64.3) | -86.0 (147.1) | -68.1 (69.8)
  4 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  4 hours post Day 1 dose | -64.9 (124.3) | -43.7 (36.1) | -26.6 (16.6) | -48.7 (77.5)
  6 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  6 hours post Day 1 dose | -68.8 (80.5) | -6.0 (73.5) | -72.9 (89.6) | -40.7 (87.0)
  9 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  9 hours post Day 1 dose | -62.8 (85.3) | -46.6 (240.7) | -84.6 (78.6) | -54.1 (93.2)
  10 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  10 hours post Day 1 dose | -7.7 (99.4) | -8.4 (114.7) | -45.0 (73.2) | -5.7 (127.9)
  11 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  11 hours post Day 1 dose | -35.6 (60.9) | -41.1 (84.5) | -70.3 (58.3) | -55.0 (113.8)
  12 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  12 hours post Day 1 dose | -49.6 (48.1) | -61.9 (88.1) | -112.1 (144.6) | -76.6 (90.3)
  14 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  14 hours post Day 1 dose | -139.0 (248.4) | -60.9 (124.3) | -99.7 (82.1) | -67.3 (63.7)
  24 hours post Day 1 dose: number analyzed (Participants) | 9 | 7 | 7 | 7
  24 hours post Day 1 dose | -115.2 (118.8) | 20.4 (252.6) | -110.4 (111.7) | -37.9 (104.5)
  Time of Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  Time of Day 7 dose | -173.1 (306.8) | -23.7 (296.2) | -150.7 (91.2) | -97.4 (176.7)
  1 hour post Day 7 dose: number analyzed (Participants) | 8 | 7 | 6 | 7
  1 hour post Day 7 dose | -101.1 (169.1) | -22.6 (63.4) | -114.7 (173.3) | -100.7 (135.0)
  2 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  2 hours post Day 7 dose | -2.9 (20.6) | -13.0 (69.7) | -88.1 (158.9) | -63.1 (86.7)
  4 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  4 hours post Day 7 dose | -78.3 (185.0) | -5.3 (98.8) | -13.4 (33.7) | -31.1 (77.4)
  6 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  6 hours post Day 7 dose | -86.4 (122.3) | 16.6 (167.4) | -57.6 (96.7) | -6.9 (122.6)
  9 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  9 hours post Day 7 dose | -100.4 (152.3) | -80.6 (211.5) | -44.3 (71.7) | -36.3 (137.6)
  10 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  10 hours post Day 7 dose | -54.9 (238.4) | -8.6 (189.4) | -7.0 (72.1) | 30.4 (176.4)
  11 hours post Day 7 dose: number analyzed (Participants) | 7 | 7 | 7 | 7
  11 hours post Day 7 dose | -37.0 (49.1) | -51.3 (106.2) | -63.0 (48.7) | -48.7 (118.8)
  12 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  12 hours post Day 7 dose | -52.3 (42.6) | -67.0 (55.5) | -128.7 (141.0) | -80.3 (97.3)
  14 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  14 hours post Day 7 dose | -141.4 (271.8) | -25.0 (21.5) | -83.0 (100.9) | -47.3 (51.2)
  24 hours post Day 7 dose: number analyzed (Participants) | 8 | 7 | 7 | 7
  24 hours post Day 7 dose | -219.8 (202.5) | 104.3 (257.0) | -199.4 (135.5) | 35.4 (66.4)

47. Secondary Outcome: Change From Baseline in 24-hour Urine Output
Description: Changes from baseline in 24-hour urine output for samples taken on Day 1 and Day 7 will be summarized by cohort. The baseline value was the last value observed prior to first administration of study drug on Day -1.
Time Frame: Baseline (Day -1), Day 1, and Day 7
Population: The PDAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan. Values were not available for all participants in the PDAS at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mL
  Day 1: number analyzed (Participants) | 9 | 7 | 7 | 7
  Day 1 | 2175.3 (2629.2) | 1794.4 (1697.0) | 3041.1 (889.2) | 1329.9 (916.7)
  Day 7: number analyzed (Participants) | 8 | 7 | 7 | 7
  Day 7 | 1995.6 (2294.0) | 1744.6 (1658.7) | 1843.6 (1027.7) | 458.4 (2233.7)

48. Secondary Outcome: Change From Baseline of the Estimated Glomerular Filtration Rate (eGFR)
Description: Changes from baseline of eGFR derived from the serum creatinine concentrations for samples taken at Day 1 (postdose), Day 2, Day 7, Day 8, and Day 35 will summarized by cohort
Time Frame: Baseline (Day 1) to end of study (35 days)
Population: The PDAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan. Of these, all 31 subjects contributed PD endpoints to the Day 1/2 assessment; 30 subjects contributed data to the Day 7/8 PD endpoints and scheduled EOS assessments.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mL/min/1.73 m²
  Day 2 | -7.4 (7.2) | -3.9 (8.8) | -2.1 (4.3) | -1.9 (3.1)
  Day 7: number analyzed (Participants) | 8 | 7 | 8 | 7
  Day 7 | -11.9 (10.0) | -3.0 (3.7) | -5.3 (3.7) | -3.4 (4.1)
  Day 8: number analyzed (Participants) | 8 | 7 | 8 | 7
  Day 8 | -9.1 (12.5) | -2.9 (3.3) | -5.5 (4.8) | -3.4 (3.5)
  Day 35: number analyzed (Participants) | 8 | 7 | 8 | 7
  Day 35 | -0.9 (8.4) | 0.0 (8.3) | 2.1 (4.3) | -3.7 (3.2)

49. Secondary Outcome: Change From Baseline in Total Kidney Volume
Description: Changes from baseline (Day -1) in total kidney volume, measured by abdominal MRI on Day 7 and Day 35, will be summarized by cohort.
Time Frame: Baseline (Day -1) to end of study (36 days)
Population: The PDAS consisted of all 31 subjects in the Safety analysis set who received lixivaptan. Overall, all 31 subjects contributed PD endpoints to the Day 1/2 assessment; 30 subjects contributed data to the Day 7/8 PD endpoints and scheduled EOS assessments; however, values were not available for all participants at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mL
  Day 7: number analyzed (Participants) | 8 | 6 | 8 | 6
  Day 7 | -8.75 (42.47) | 4.97 (30.84) | -66.19 (141.47) | 23.58 (33.69)
  Day 35: number analyzed (Participants) | 8 | 5 | 8 | 6
  Day 35 | -26.63 (77.84) | -3.78 (26.06) | -4.29 (81.27) | 28.88 (68.16)

50. Secondary Outcome: Change From Baseline in Liver Volume
Description: Changes from baseline (Day -1) in liver volume, measured by abdominal MRI on Day 7 and Day 35, will be summarized by cohort.
Time Frame: Baseline (Day -1) to end of study (36 days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mL
  Day 7: number analyzed (Participants) | 8 | 6 | 8 | 6
  Day 7 | 53.04 (125.51) | 43.02 (92.15) | 104.01 (131.21) | -0.03 (40.98)
  Day 35: number analyzed (Participants) | 8 | 5 | 8 | 6
  Day 35 | -6.70 (86.74) | 28.66 (99.77) | 53.51 (82.52) | -11.00 (109.04)

51. Secondary Outcome: Change From Baseline of Plasma Copeptin
Description: Changes from baseline (Day -1) in plasma copeptin, a marker for circulating vasopressin, at Day 2, Day 7, and Day 35 will be summarized by cohort.
Time Frame: Baseline (Day -1) to end of study (36 days)
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
pmol/L
  Day 2 | 5.072 (4.798) | 1.986 (3.286) | 12.655 (15.527) | -1.986 (10.893)
  Day 7: number analyzed (Participants) | 8 | 7 | 8 | 7
  Day 7 | 9.745 (4.910) | 3.016 (3.392) | 17.906 (10.321) | 34.519 (89.262)
  Day 35: number analyzed (Participants) | 8 | 7 | 8 | 7
  Day 35 | 2.111 (2.829) | 2.786 (5.498) | -0.943 (8.435) | -3.337 (13.993)

52. Secondary Outcome: Change From Baseline in Serum Creatinine
Description: Changes from baseline in serum creatinine for samples taken at Day 2, Day 7, Day 8, and Day 35 will be summarized by cohort.
Time Frame: Baseline (Day 1, predose) to end of study (35 days)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
umol/L
  Day 2 | 6.7778 (6.13958) | 4.1429 (7.17469) | 4.7500 (13.49868) | 4.5714 (5.62308)
  Day 7 | 12.6667 (9.73396) | 2.7143 (3.45033) | 19.2500 (16.88406) | 6.5714 (8.86674)
  Day 8 | 11.1111 (11.94199) | 2.2857 (3.14718) | 17.6250 (12.81670) | 7.5714 (7.48013)
  Day 35 | 2.4004 (6.87657) | 0.8571 (6.59365) | -8.5000 (14.04076) | 7.5714 (5.12696)

53. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN)
Description: Changes from baseline in BUN for samples taken at Day 2, Day 7, Day 8, and Day 35 will be summarized by cohort.
Time Frame: Baseline (Day 1, predose) to end of study (35 days)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 9 | 7 | 8 | 7
mmol/L
  Day 2 | 0.0644 (0.82257) | -0.1743 (0.43535) | -0.1563 (1.15821) | -0.1300 (1.16973)
  Day 7 | -0.2000 (1.17573) | -0.0614 (1.29029) | -0.7488 (1.66207) | 0.2014 (1.59194)
  Day 8 | -0.5711 (1.14740) | -0.1043 (1.22296) | -0.2338 (1.43097) | -0.1229 (0.99856)
  Day 35 | 0.0008 (1.61696) | -0.1886 (1.36772) | -0.2338 (2.08729) | 0.2286 (1.94233)

54. Other Pre Specified Outcome: Volume of Distribution Over 24 Hours After Extravascular Dosing (VZ/F24H) of Lixivaptan in ADPKD Patients
Description: The pharmacokinetic parameter VZ/F24H for lixivaptan, calculated as CL/F24H divided by Day 7 PM λZ, will be summarized by cohort. VZ/F24H was not specified in the statistical analysis plan and was calculated for the combined 24-hour period including AM and PM dosing intervals on Day 7. This parameter replaces VZ/F initially planned for the Day 7 AM dose.
Time Frame: Day 7 (am)
Population: Of the 31 subjects in the PKAS, 29 contributed data to Day 7 (am). Data were excluded for 1 subject in the low dose/CKD1 or 2 cohort from Day 1 (pm) onwards due to substantial deviations from planned dosing interval durations. Missing values and substantial deviations meant additional results were excluded from subjects at various time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 6 | 4 | 7 | 6
L | 547.4 (57.4) | 546.0 (48.2) | 515.1 (50.7) | 731.8 (38.4)

55. Primary Outcome: Aquaretic Tolerability of Lixivaptan Measured by a Tolerability Questionnaire Relating to the Symptom Burden of Nocturia, Urgency, and Frequency at Day 7: Question 7
Description: The number of study participants who answered "not at all" and "slightly" to the following question at Day 7 will be measured:
  • If the study drug made you go to the bathroom (urinate) more often than usual during the night, did it bother you?
Time Frame: Day 7
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Lixivaptan / CKD1 or CKD2; Low Dose Lixivaptan / CKD1 or CKD2; High Dose Lixivaptan / CKD3; Low Dose Lixivaptan / CKD3: Oral low dose lixivaptan in participants with CKD3
  Lixivaptan: Oral vasopressin V2 receptor antagonist
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
Number analyzed (Participants) | 6 | 3 | 6 | 4
Participants
  Answered "not at all" | 2 | 1 | 2 | 1
  Answered "slightly" | 3 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | High Dose Lixivaptan / CKD1 or CKD2 | Low Dose Lixivaptan / CKD1 or CKD2 | High Dose Lixivaptan / CKD3 | Low Dose Lixivaptan / CKD3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/9 | 4/7 | 4/8 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Lixivaptan / CKD1 or CKD2 (N=9) | Low Dose Lixivaptan / CKD1 or CKD2 (N=7) | High Dose Lixivaptan / CKD3 (N=8) | Low Dose Lixivaptan / CKD3 (N=7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03487913/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT03487913/SAP_001.pdf